CLINICAL TRIAL: NCT04249271
Title: Antithyroidale Antikörper Mit Oder Ohne Subklinische Hypothyreose Bei Weiblicher Infertilität in Der Schwangerschaft Und im Wochenbett.
Brief Title: Antithyroidal Antibodies With or Without Subclinical Hypothyroidism During Pregnancy in Infertile Women
Acronym: Anti-TPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christian De Geyter, Prof., University Hospital, Basel, Switzerland
Other Study IDs: EKNZ 39-009 00960
Record Dates: First submitted 2018-02-17; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Thyroid Gland Disease; Pregnancy Complications
Keywords: thyroid; antibody; pregnancy; infertility
MeSH Terms: conditions — Thyroid Diseases; Pregnancy Complications; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- euthyroid, no antibodies: TSH 0.3 to 2.5 mIU/l and anti-TPO <100 IU/ml repeated serum sampling
  Interventions: Other: serum sampling
- borderline euthyroid, no antibodies: TSH 2.5 to 4.5 mIU/l and anti-TPO <100 IU/l repeated serum sampling
  Interventions: Other: serum sampling
- hypothyroidism, no antibodies: TSH >4.5 mIU/l and anti-TPO <100 IU/ml repeated serum sampling
  Interventions: Other: serum sampling
- euthyroid, with antibodies: TSH 0.3 to 2.5 mIU/l and anti-TPO >100 IU/ml repeated serum sampling
  Interventions: Other: serum sampling
- borderline euthyroid, with antibodies: TSH 2.5 to 4.5 mIU/l and anti-TPO >100 IU/l repeated serum sampling
  Interventions: Other: serum sampling
- hypothyroidism, with antibodiesal: TSH >4.5 mIU/l and anti-TPO >100 IU/ml repeated serum sampling
  Interventions: Other: serum sampling

INTERVENTIONS:
Other: serum sampling — repeated serum sampling during pregnancy and thereafter

SUMMARY:
One prospective observational study was carried out in 2009 aiming at identifying the fluctuations of the thyroid hormones in women with normal thyroid gland and in women with anti-TPO antibodies. Serum samples were collected periodically during and after pregnancy in previously infertile women. The samples were stored frozen at -80 °C. Now, the hormone measurements will be carried out.

DETAILED DESCRIPTION:
Exclusion of thyroid disease has long been an integral part of a comprehensive infertility work-up, because thyroid function disorders are also associated with disturbances in the menstrual cycle and can cause complications during pregnancy. Subclinical hypothyroidism is the most frequent disease of the thyroid in women of reproductive age (affecting 5 to 10 %). For a long time, measurement of TSH concentration was the only screening parameter used to exclude thyroid disorders. Not only has the differentiation of normal thyroid function (euthyroidism) from the pathological range been controversial for some years but, recently, the role of an elevated anti-TPO antibody titre has also been identified as a significant and independent risk factor for miscarriages and for complications during late pregnancy, even in otherwise euthyroid women. This discovery implies that solely determining the TSH concentration is insufficient. The mechanism underlying the increased rate of complications during pregnancy is also unclear.

The investigators therefore performed a double study to clarify the relative importance of the various possible parameters of thyroid function in the context of an infertility work-up:

1. Prevalence study: Measurement of TSH and anti-TPO concentrations in 175 women who present with infertility at the Infertility Clinic at the Women's Hospital, University Hospital Basel. In addition, each participant underwent an ultrasound scan of the thyroid. Control group: 175 healthy women of reproductive age and with regular menstrual cycles, but not currently wishing to have children (recruited via posters in the university and Blood Donor Centre). This study has been finished in 2010. The data of the prevalence study were used to carry out the prospective sampling of the serum samples.
2. Prospective measurement of fluctuations in thyroid function during pregnancy and post-partum in a group of euthyroid women and/or those with subclinical hypothyroidism (TSH > 4.5 mIU/l) with/without anti-TPO antibodies. Two different euthyroid groups were defined for the study: Euthyroidism I = TSH 0.3-2.5 mIU/l; Euthyroidism II = TSH 2.5-4.5 mIU/l. Six groups, each with 16 women, divided according to TSH concentration and anti-TPO antibody status, will be required (total 96). All female participants with subclinical hypothyroidism (TSH concentration > 4.5 mIU/l, normal values of peripheral thyroid hormones) receive a T4 supplementation dose. Serum samples will be collected each week from the start of pregnancy up to the 12th week and stored frozen at -80 °C. Thereafter, a serum sample will be collected once a month (up to the 38th week) and stored frozen at -80 °C. Finally, one serum sample post-partum (4 to 6 weeks after delivery) and freeze it. A total of 96 women (16 in each group) were recruited to participate in this study.

After conclusion of the observation period, levels of the following hormones will be measured in the total of 1120 serum samples: TSH, total and free l-thyroxine and fT4 index, total and free triiodothyronine, thyroid autoantibodies (TPO antibodies), hCG, 17β-oestradiol, progesterone, prolactin.

ELIGIBILITY:
Inclusion Criteria:

* previous infertility with known thyroidal function (TSH, anti-TPO)

Exclusion Criteria:

* other endocrine pathology, such as Addison, diabetes mellitus
* manifest thyroidal pathology, such as Graves disease
* contraindication against pregnancy
* after repeated miscarriage (3 or more)
* heavy smokers (20 cig per day or more)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy after infertility
Study Population: Healthy women having become pregnancy after infertility.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Deviations from euthyroid function as given by serum levels of TSH (expressed in mIU/l) during pregnancy and after birth. | 12 months
  Impact of antibodies on thyroid function during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geyter, Prof., Principal Investigator — University of Basel
Locations (1):
- Klinik für Gyn. Endokrinologie und Reproduktionsmedizin der Frauenklinik des Universitätsspitals, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
The serum samples are coded and cannot be traced back to individual patients.